CLINICAL TRIAL: NCT06039436
Title: Conditioning Regimen Containing Low Dose ATG for The Treatment of Acquired Severe Aplastic Aplasia Receiving Single Cord Blood Transplant: A Multi-center, Single-arm Study
Brief Title: Conditioning Regimen Containing Low Dose ATG for The Treatment of Acquired SAA Receiving sUCBT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Xiaoyu Zhu, Chief physician, Anhui Provincial Hospital
Other Study IDs: CBSAA001
Record Dates: First submitted 2023-09-09; First posted 2023-09-15 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Severe Aplastic Anemia
Keywords: Anti-Thymocyte Globulin (Rabbit); Umbilical Cord Blood Transplantation; Severe Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic | interventions — Antilymphocyte Serum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ATG group: Patients in the ATG group will be treated with conditioning regimen containing ATG 2mg/kg on day -7 prior to transplant.
  Interventions: Drug: Anti-Thymocyte Globulin (Rabbit)

INTERVENTIONS:
Drug: Anti-Thymocyte Globulin (Rabbit) — Indications for trial stopping: subjects occur pregnancy events, severe organ function impairments, or emergency events related or unrelated to treatment; or subjects are unwilling to continue participating in the clinical trial.

SUMMARY:
To evaluate the safety and efficacy of Single Umbilical Cord blood transplantation (sUCBT) containing low dose ATG based conditioning regimen in the treatment of acquired Severe Aplastic Anemia (SAA).

DETAILED DESCRIPTION:
Hematopoietic stem cell transplantation (HSCT) from HLA-compatible sibling donors is the standard preferred therapy for Severe Aplastic Anemia (SAA). At present, HLA-compatible donors in China fail to meet the needs of patients for transplantation. Umbilical Cord blood transplantation (UCBT) is an alternative treatment for patients with emergency conditions who lack compatible sibling donors, have failed immunosuppressant therapies or cannot wait for unrelated fully compatible donors. However, implantation failure is one of the main problems in UCBT for SAA due to the low cord blood stem cells. Nowadays, there is no consensus on the optimal conditioning regimen for UCBT treatment of SAA, and whether ATG should be added to the conditioning regimen is still controversial. Early clinical studies in UCBT have shown that the sufficient ATG in the conditioning regimen will lead to a decrease rate of implantation rate and affect survival of UCBT ultimately. However, a range of recent studies have found that with the addition of low-dose ATG, T cell reconstitution seems to outperform bone marrow or peripheral blood stem cell transplantation. Therefore, how to properly use ATG to both retain its effective GVHD prevention effect and reduce its impact on immune reconstruction has important clinical significance for improving the transplantation efficacy. In this study, a multicenter clinical study will be conducted to observe the safety and efficacy of UCBT with low dose ATG in the treatment of SAA and the long-term quality of life of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with severe aplastic anemia who do not respond to initial diagnosis or immunosuppressive therapy;
* Patients meet diagnostic criteria for severe aplastic anemia (Camitta criteria);
* Age from 1 to 50 years old, male or female;
* Patients without HLA-matched sibling or unrelated donors avaliable;
* Patients who have undergone unrelated cord blood transplantation need to have HLA high-resolution matching、TNC (before cord blood freezing)≥3.0×107/kg、CD34+(before cord blood freezing)≥1.5×107/kg、tubule recovery rate≥80%;
* patients and their family members or guardians agreed to the study and signed informed consent;
* No severe organ failure;
* ECOG score≤2 and HCT-CI≤2;
* serum ferritin (SF)<1000ug/L;
* women of reproductive agemust have a negative pregnancy test and agree to use effective contraception during treatment and for one year thereafter.

Exclusion Criteria:

* patients with inherited bone marrow failure syndromes;
* Positive for HLA-A, B, Cw, DRB1, DQB1, DPB1 site-specific HLA antibodies for donor cord blood with solid-phase fluorescence assay;
* patients who have previously received allogeneic hematopoietic stem cell transplantation or solid organ transplantation;
* Uncontrolled bacterial, viral, or fungal infections;
* HIV infection or active viral hepatitis B or C infection;
* Pregnant or breastfeeding women;
* patients with a history of primary malignancy within 3 years prior to transplant treatment;
* patients receiving ATG treatment within 2 weeks before transplantation;
* patients with drug dependent or uncontrolled mental illness or cognitive impairment;
* Participants in other similar clinical studies within 3 months;
* Patients allergic to ATG;
* patients considered unsuitable for inclusion by the researchers.

Ages: 1 Year to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients with indications for hematopoietic stem cell transplantation and initially diagnosed with severe aplastic anemia or have not responded to immunosuppressive therapy
Sampling Method: Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
The one-year probability of GRFS | one year
  GRFS is defined as survival without grade III-IV acute GVHD immunosuppression requiring chronic GVHD or relapse.

SECONDARY OUTCOMES:
The cumulative incidence of platelet engraftment at 28 days after transplantation | 28 days
  Platelet engraftment is defined as independent from platelet transfusion for at least 7 days with a platelet count of more than 20 × 10^9/L.
The cumulative incidence of neutrophil engraftment at 28 days after transplantation | 28 days
  Neutrophil engraftment is defined as neutrophil count achieves 0.5 ×10^9/L for three consecutive days.
Time of platelet engraftment | 28 days
  Platelet engraftment is defined as independent from platelet transfusion for at least 7 days with a platelet count of more than 20 × 10^9/L.
Time of neutrophil engraftment | 28 days
  Neutrophil engraftment is defined as neutrophil count achieves 0.5 ×10^9/L for three consecutive days.
The cumulative incidence of acute GVHD at 100 days after transplantation | 100 days
  Acute GVHD is defined that occurs within 100 days after transplantation
The cumulative incidence of chronic GVHD at 100 days after transplantation | one year
  Chronic GVHD is defined that occurs 100 days after transplantation
Immune reconstitution after transplantation | one year
  The level of immunoglobulin, T cells, B cells and NK cells reconstitution after transplantation
The 180-day probability of TRM | 180 days
  TRM(transplant-related mortality) is defined that death due to any transplant-related cause within 180 days after transplantation
The incidence of infection | one year
  Infection is defined as various post-transplant associated infections
The one-year probability of OS | one year
  OS (overall survival) is defined as the time which begins at diagnosis and up to the time of death
The one-year probability of DFS | one year
  DFS (disease free survival) is defined as the time from treatment until the recurrence of disease (or death) after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyu Zhu, ph.D, Principal Investigator — The First Affiliated Hospital of University of Science and Technology of China (Anhui Provicial Hospital)
Locations (1):
- The First Affiliated Hospital of University of Science and Technology of China (Anhui Provincial Hospital), Hefei, Anhui, China